CLINICAL TRIAL: NCT06291480
Title: Music Therapy After Stroke (Subacute Phase): Assessing the Impact of Motivation and Neuroplasticity on Recovery of Upper-limb Impairment and Attention Deficits
Brief Title: Music Therapy After Stroke (Subacute Phase)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient inclusions in the available time after an extension of 50% with the sample at 16/20.
Sponsor: Universiteit Leiden (Other)
Collaborators: Amstelring (Unknown)
Responsible Party: Principal Investigator, Rebecca Schaefer, Associate professor, Universiteit Leiden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL78853.058.22 / STRUM
Record Dates: First submitted 2024-02-07; First posted 2024-03-04 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Stroke (CVA) or TIA; Stroke/Brain Attack
Keywords: Music Therapy; Neurologic Music Therapy; Movement rehabilitation; Cognitive rehabilitation; Motivation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Intervention period compared to care as usual in cross-over design.
Who Masked: Outcomes Assessor
Masking Description: Analyses will be done after blinding to participant id and gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy + Care as Usual (Experimental): 9 music therapy sessions within 2-5 weeks during stroke rehabilitation, in addition to care as usual.
  Interventions: Behavioral: Neurologic Music Therapy
- Care as Usual (No Intervention): 2-5 weeks of care as usual, without music therapy

INTERVENTIONS:
Behavioral: Neurologic Music Therapy — Music therapy focused on cognitive and motor rehabilitation after stroke (subacute phase).
  Arms: Music Therapy + Care as Usual

SUMMARY:
The goal of this longitudinal, single-subject study is to investigate the role of motivation in music therapy for stroke patients within the subacute phase, who experience upper limb and/or attention deficits. The main questions it aims to answer are:

* Does music therapy increase patient's motivation to rehabilitate?
* Do increases in motivation correlate with functional improvements, in particular upper limb and/or attention skills?

Participants will receive up to 9 music therapy sessions within 3-5 weeks, with functional assessments before and after each period. Each participant serves as their own comparison: researchers will compare a period with standard care only (control phase) to a period with music therapy plus standard care (intervention phase), the order of which will be randomized in advance.

DETAILED DESCRIPTION:
Rationale: Stroke is a highly disabling condition, for which music therapy is regularly used in rehabilitation. Motivation is considered to be a mechanism for functional improvements, including in neurologic music therapy (NMT), likely due to potential mood improvements, but it is not generally explicitly investigated. This motivation level may in turn affect not only functional outcomes and subjective well-being, but also adherence to other rehabilitation therapies.

Objectives: The primary goal of the study is to investigate motivation as an underlying mechanism of neurologic music therapy (NMT) for stroke patients experiencing upper-limb impairments and/or cognitive deficits, in the sub-acute phase of stroke. A secondary goal is to assess NMT-related changes in motor function, cognitive outcomes, and self-reported measures of well-being.

The hypothesis is that NMT will increase motivation, and that increased motivational state will positively affect functioning in both motor and/or cognitive domains.

Study design: The study has a longitudinal, single-subject design; as stroke patients are not a homogenous group, this design is adopted to control for expected within-subject variations. To account for variability in brain damage that is caused by stroke, each subject thus serves as their own control, and a longitudinal, repeated-measures design is selected. Participants will be randomized into two groups for a cross-over design, either receiving the intervention or the control phase first or vice versa, which counters order effects and assesses intervention effectiveness (as part of the secondary goals).

All subjects will receive NMT targeting both upper- limb movement and attention. All participants will receive a target of 9 NMT sessions (participants who complete a minimum of 6 sessions will be included in the analysis) over 3-6 weeks (depending on the rehabilitation trajectory, as subacute patients generally are admitted for a minimum of ± 6 and a maximum of 16 weeks), aiming for an average of 3 sessions per week, but adjusted to a patient's expected length of stay and ability, using a tailored approach.

Participants will receive three measurements. A baseline measure (TP1), on the first week of the rehabilitation trajectory, a second measure (TP2) either after the treatment/intervention period or control/ care as usual period (depending on the randomisation) and a post-treatment (TP3). The time interval between TP1- TP2 and TP2-TP3 are at least 21 days (3 weeks), with a margin of maximum 4-7 days, depending on their expected length of stay in the care facility.

Study population: In order to be eligible to participate in the study, a participant should be above 18 years of age and have had their first-ever supratentorial stroke between 2 weeks and up to 6 months before enrollment. Moreover, participants will have a referral for a paretic upper limb, i.e., partial loss of the capacity to carry out a voluntary upper limb movement and/or difficulty with attention/concentration, (e.g., complaints of being easily distractible, or unable to focus on a specific task in the presence of competing information, or complain of decline in attention). Participants must be able to receive music therapy for a minimum of 2-3 sessions per week, aiming for a total of 9 sessions over a minimum of three weeks, reducing this to 6 sessions in 2 weeks if required. The frequency of sessions is based on their ability and expected length of stay. Good command of the Dutch or English language is also a prerequisite for participation.

Participants will be excluded if this is not their first stroke or if a second stroke occurs during their stay. Further exclusion criteria are the following: i) upper limb paralysis as assessed by a score < 2 points on the Medical Research Scale (MRC) for muscle strength; ii) severe behavioural and/or cognitive problems preventing understanding or carrying out instructions or risk of dementia (a score <21 on the Mini-mental state examination; MMSE); iii) severe communication problems, e.g., severe aphasia and/or apraxia of speech; iv) known psychiatric, substance abuse, or neurological comorbidity. For participants who score <24 on the MMSE, a follow-up check will be carried out for a possible dementia diagnosis which would retrospectively lead to exclusion.

Sample size: In a previous study, 40 stroke patients in the sub-acute phase were allocated to either twenty 30-minute sessions of music-supported therapy (N = 20; 4 withdrew/excluded; 16 in final analysis) or twenty additional sessions of conventional therapy (N = 20; 2 withdrew/excluded; 18 in final analysis). The study found a significant correlation (r = .562, p = .024) between patients' intrinsic motivation to engage in musical activities as measured by the BMRQ at baseline and improvement of upper-limb function as measured by the Action Research Arm Test (ARAT) at 3 months, which was not found in the comparator of occupational/physical therapy (r = -.305, p < .21), with a significant difference between correlations (z = 2.4, p < .05). Using G power 3 analysis, the investigators estimated that 18 participants are needed to observe a similar effect size for a sufficiently powered study (α=0.05 and (1-β)=0.8; ρ H1 = 0.56). This indicates that 20 participants completing the entire protocol would be required to observe an effect of motivation in music therapy, with an expected attrition/missing data rate of 10-20%. This sample size is similar to the number of participants used in studies showing an effect for our secondary objectives, ranging from 14-20 participants, on the effects of music therapy on motor function, cognition, and psychological wellbeing. Recruitment will continue until 20 participants have completed the protocol.

Intervention: The intervention condition will consist of a target of up to 9 sessions in total, administered over an average of 5 weeks, but may span from 2 to 8 weeks according to the patient's length of stay at the Leo Polak Stroke Rehabilitation Centre. All music therapy interventions will be delivered by a registered music therapist. The protocol aims for participants to receive a minimum of two sessions per week over the duration of the study enrollment. However, this schedule may not be possible in every case due to the participants' length of stay. Participants who complete a minimum of 6 sessions will be included in the final analyses. The number of sessions each participant receives will be recorded and treated as a variable systematically recorded, and the number of sessions will be accounted for in the statistical analysis.

Main parameters/ endpoints: The main parameters of the study focus on the differences in motivation levels of participants as the result of applying NMT techniques in the subacute phase of stroke, comparing within-subject differences between changes related to the intervention and the control period. The motivation level of participants will be measured using the BMQ-S [patient-rated] as state-level motivation. The secondary parameters relate to behavioural outcomes of upper limb, and cognitive functions, as well as self-reported measures of well-being following NMT for within-participant comparisons between the intervention and control period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had their first-ever supratentorial stroke between 2 weeks and up to 6 months before enrolment
* Paretic upper limb and/or attention/ concentration problems
* Ability to communicate in Dutch or English

Exclusion Criteria:

* Severe (global) aphasia
* paralysis of upper limb
* severe cognitive decline (MMSE <24)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Motivation: Brain Injury Rehabilitation Trust Motivation Questionnaire (BMQ-S) [self-reported] | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The BMQ-S is a 34-item questionnaire, which measures the motivation levels of the stroke survivor, using a 4-point likert scale (always, often, sometimes, never). Items that involve different factors such as anhedonia, perseveration, poor initiation, or distractibility, are summed to create a total score from 34 to 136, with higher scores representing greater difficulties in motivation.

SECONDARY OUTCOMES:
Motor Function: Action Research Arm Test (ARAT) | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The Action Research Arm Test (ARAT) is a 19-item observational measure used by healthcare professionals to assess upper extremity performance (coordination, dexterity, and functioning) in stroke recovery and brain injury. Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch, and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Performance on each item is rated on a 4-point ordinal scale ranging from:
  3) Performs test normally 2) Completes test, but takes abnormally long or has great difficulty
  1) Performs test partially 0) Can perform no part of test
  The maximum score on the ARAT is 57 points (possible range 0 to 57). A higher score indicates better functioning in the upper extremity.
Motor Function: Barthel Index (BI) | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.
  The ten items are scored on a 4/5-item Likert scale, and then a final score is calculated by summing the points awarded to each functional skill. This allows the examiner to measure a patient's functional disability by quantifying their performance.
  Minimum value: 0, maximum value: 20. The higher the score, the more independent the patient is in completing the measured ADLs. Higher scores also indicate the patient is more likely to return home, with varying degrees of assistance, following hospital discharge. The lower the score, the more dependent the patient is with ADL completion.
Cognition: Cancellation Wechsler Adult Intelligence Scale (WAIS-IV) | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The WAIS-IV cancellation test measures, amongst others, processing speed, visuospatial attention and/or neglect. A score is constructed based on how many targets or false alarms are indicated within 45s. More missed targets or false alarms indicate worse performance.
  The test does not explicitly list minimum or maximum scores due to the nature of the test being a scaled score rather than a fixed value. However, based on the understanding that scaled scores typically range from 1 to 19, with lower scores indicating more cognitive difficulties and higher scores indicating fewer difficulties, investigators infer that the lowest possible scaled score would be around 1, and the highest possible scaled score would be around 19. This is assuming that the test follows typical scoring conventions where the mean is approximately 10 and the standard deviation is about 3
Cognition: Color-Word Interference Test, also known as Stroop test | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The Stroop test can be used to measure a person's processing speed and interference, testing overall executive processing abilities. It is based on the difference of reading and naming ink colors of a word name when the name and color are different than when they are the same.
  The interference is calculated by subtracting congruent trials (only naming colors or words) with interference trials (words printed in colored ink), taking into account mistakes, with less difference in time o fewer mistakes indicating better performance.
Cognition: WAIS IV Digit Span Test - Forward and Backward | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The Digit Sequencing or Digit Span test is one of the main tools developed to measure one's working memory and attention.
  The Digit Span score is the length of the longest correctly repeated sequence, either forward or backward. The number of sequences of correctly recalled digits is summed to produce a raw score between 0 and 8 for each subtest, where a higher score indicates better performance.
Cognition: Verbal Fluency Test | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  A verbal fluency test is a kind of test in which a participant is asked to produce as many words as possible from a category in a given time (usually 60 seconds).
  The phonemic verbal fluency test consists of producing as many words as possible within one minute for 3 letters (using cross-validated versions that are different at each time point). The total number of valid responses across trials excluding repeats are added to produce a total score, where a higher score indicates better performance.
Cognition: Trail Making Test (TMT) | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The trail making test assesses a wide variety of cognitive processes including attention, visual search and scanning, sequencing and shifting, psychomotor speed, abstraction, flexibility, ability to execute and modify a plan of action, and ability to switch instructions.
  The Trail Making Test is measured in time over 5 trials. The final score is trial 2 (number/letter-switching) trial 1 (only using numbers). The interference is scored based on the difference between trials 1 and 2, where a larger time difference indicates more interference.

OTHER OUTCOMES:
Motivation to engage in musical activities: Barcelona Music Reward Questionnaire (BMRQ) | This outcome measure will be administered once, during the baseline Test Point (TP1) (week 1).
  The BMRQ measures intrinsic motivation to engage in musical activities and experience musical reward. The BMRQ examines five main facets that characterize musical reward experience in individuals: musical seeking, emotion evocation, mood regulation, social reward, and sensory-motor.
  The BMRQ is a 20-item questionnaire in which participants rate on a 5-point scale the extent to which they agree with statements indicating their degree of musical reward across five dimensions: musical seeking, emotion evocation, mood regulation, sensory-motor, and social reward. Scores are constructed by summing the likert scale score, ranging from 20-100.
Quality of Life: EuroQol-5 (EQ-5D-5L) | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The EQ-5D-5L is an outcome measure for measuring the health and health-related quality of life, assessing five important dimensions: mobility, self-care, daily activities, pain and fear/depression (5D) represented in 5 questions. Score range from 1-5 per question where a higher number is a worse outcome (score range between 1 and 25), and a visual analogue scale from 0-100 where for both a higher number is a better outcome.
Mood: Depression Anxiety Stress Scale-21 (DASS-21) | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Scores of the Depression Anxiety Stress Scale are added up per category (depression, anxiety and stress):
  Depression symptoms related items: 3, 5, 10, 13, 16, 17, 21 (range from 0-21) Anxiety disorder-related items: 2, 4, 7, 9, 15, 19, 20 (range from 0-21) Stress-related items: 1, 6, 8, 11, 12, 14, 18 (range from 0-21), where a higher score indicates a worse outcome for all domains.
Mood: Visual Analogue Mood Scale (VAMS) | Within 10 minutes before the start of each music therapy session (pre intervention) and immediately after each music therapy session (post intervention).
  The VAMS consists of a 180-mm line having two circles at its respective ends that represent two opposite moods - the upper circle containing a stylized "happy" face, the lower a "sad" one. The VAMS thus allows measuring euthymia/dysthymia along a continuum. Scores are measured by locating responses on the line (min 0 - max 180).
Personality Traits: The Big Five Index-Extra Short Form (BFI-2-XS) | This outcome measure will be administered once, during the baseline Test Point (TP1) (week 1).
  The BFI-2 is a measure of the Big Five personality domains (labelled as Extraversion, Agreeableness, Conscientiousness, Negative Emotionality, and Open-Mindedness) through 15 more specific question items that are scored on a Likert scale from 1-5 and combined per personality domain (score range is 3-15 per domain).
  Higher scores indicate a greater tendency toward that personality trait (e.g., higher values of Conscientiousness indicate propensity to orderliness, industriousness, and dutifulness, whereas higher values of Negative Emotionality indicate propensity to anxiety, depression, and lability).
Optimism: Life Orientation Test- Revised (LOT-R) | This outcome measure will be administered once, during the baseline Test Point (TP1) (week 1).
  The LOT-R will be used to assess dispositional optimism. The 10-item LOT-R comprises a combination of direct scored, reverse-scored and filler items. All items are presented on 5-point scales, from 0 (I disagree a lot) to 4 (I agree a lot).
  Scores can range from 0-24, interpreted in categories, namely: 0-13: Low Optimism (High Pessimism); 14-18: Moderate Optimism; 19-24: High Optimism (Low Pessimism).
Brief self-report of therapy expectations and satisfaction with treatment | This outcome measure will be administered at 3 different time points (TP): Baseline/TP1 (week1), Mid-Trial/TP2 (week 4) and Final Measures/TP3 (week 7).
  Brief questionnaire targeting the expectations of the participant regarding music therapy, but also other disciplines, such as physical therapy, psychology, occupational therapy, etc A likert-scale is used to indicate the expectations of the participant, from 0 (totally disagree) to 4 (totally agree), with the higher scores indicating that the patient expects that a particular discipline will/will not help them improve/ rehabilitate optimally.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Hulst, PhD, Study Chair — Leiden University
Locations (1):
- Leo Polak Rehabilitation centre, Amsterdam, Nederland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
To the extent that participants give permission to share their data, Data relating to the main outcomes will be shared in online repository. Coded data will be published in an online scientific archive for the purpose of future research, in line with Open Science practices, and for the verification of findings for 10 years according to the Data Management Guidelines of the Health, Medical, and Neuropsychology Unit (v171220), Institute of Psychology, Faculty of Social and Behavioural Sciences at Leiden University. These data would not be traceable as they are not linked in any way to personal data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Coded data will be published in online scientific archive without a time limit, all participant data, including physical documents will be archived at Faculty of Social and Behavioural Sciences at Leiden university for 10 years.
Access Criteria: Coded data that cannot be traceable to the participant identifying information will be published in an online repository, the web address of the repository will be included for each publication that results from the study. No restriction to access the publicly available data will be imposed, however, future studies that use the data of the study will be required to make reference to the study AND/OR the repository.

REFERENCES:
- [Background] Altenmuller E, Marco-Pallares J, Munte TF, Schneider S. Neural reorganization underlies improvement in stroke-induced motor dysfunction by music-supported therapy. Ann N Y Acad Sci. 2009 Jul;1169:395-405. doi: 10.1111/j.1749-6632.2009.04580.x. PMID 19673814
- [Background] Baltazar, M., Västfjäll, D., Asutay, E., Koppel, L., & Saarikallio, S. (2019). Is it me or the music? Stress reduction and the role of regulation strategies and music. Music & Science, 2. https://doi.org/10.1177/2059204319844161
- [Background] Barker-Collo SL, Feigin VL, Lawes CM, Parag V, Senior H, Rodgers A. Reducing attention deficits after stroke using attention process training: a randomized controlled trial. Stroke. 2009 Oct;40(10):3293-8. doi: 10.1161/STROKEAHA.109.558239. Epub 2009 Jul 23. PMID 19628801
- [Background] Burger B, Thompson MR, Luck G, Saarikallio S, Toiviainen P. Influences of rhythm- and timbre-related musical features on characteristics of music-induced movement. Front Psychol. 2013 Apr 12;4:183. doi: 10.3389/fpsyg.2013.00183. eCollection 2013. PMID 23641220
- [Background] Dimitriadis T, Della Porta D, Perschl J, Evers AWM, Magee WL, Schaefer RS. Motivation and music interventions in adults: A systematic review. Neuropsychol Rehabil. 2024 Jun;34(5):649-678. doi: 10.1080/09602011.2023.2224033. Epub 2023 Jun 21. PMID 37340969
- [Background] Dwan T, Ownsworth T. The Big Five personality factors and psychological well-being following stroke: a systematic review. Disabil Rehabil. 2019 May;41(10):1119-1130. doi: 10.1080/09638288.2017.1419382. Epub 2017 Dec 22. PMID 29272953
- [Background] Fine, E. & Delis, D. (2011) Delis-Kaplan Executive Functioning System. In J. S. Kreutzer, J. DeLuca, and B. Caplan (Eds) Encyclopedia of Clinical Neuropsychology,. New York, NY: Springer, pp. 796-801. doi: 10.1007/978-0-387-79948- 3_1539.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Fujioka T, Dawson DR, Wright R, Honjo K, Chen JL, Chen JJ, Black SE, Stuss DT, Ross B. The effects of music-supported therapy on motor, cognitive, and psychosocial functions in chronic stroke. Ann N Y Acad Sci. 2018 May 24. doi: 10.1111/nyas.13706. Online ahead of print. PMID 29797585
- [Background] Grau-Sanchez J, Duarte E, Ramos-Escobar N, Sierpowska J, Rueda N, Redon S, Veciana de Las Heras M, Pedro J, Sarkamo T, Rodriguez-Fornells A. Music-supported therapy in the rehabilitation of subacute stroke patients: a randomized controlled trial. Ann N Y Acad Sci. 2018 Apr 1. doi: 10.1111/nyas.13590. Online ahead of print. PMID 29607506
- [Background] Grau-Sanchez J, Munte TF, Altenmuller E, Duarte E, Rodriguez-Fornells A. Potential benefits of music playing in stroke upper limb motor rehabilitation. Neurosci Biobehav Rev. 2020 May;112:585-599. doi: 10.1016/j.neubiorev.2020.02.027. Epub 2020 Feb 21. PMID 32092314
- [Background] Kim SY, Kim JM, Stewart R, Kang HJ, Kim SW, Shin IS, Park MS, Cho KH, Yoon JS. Influences of personality traits on quality of life after stroke. Eur Neurol. 2013;69(3):185-92. doi: 10.1159/000345699. Epub 2013 Jan 10. PMID 23306809
- [Background] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Background] Mas-Herrero, E., Marco-Pallares, J., Lorenzo-Seva, U., Zatorre, R. J., & Rodriguez-Fornells, A. (2012). Individual differences in music reward experiences. Music Perception: An Interdisciplinary Journal, 31(2), 118-138.
- [Background] Oddy M, Cattran C, Wood R. The development of a measure of motivational changes following acquired brain injury. J Clin Exp Neuropsychol. 2008 Jul;30(5):568-75. doi: 10.1080/13803390701555598. PMID 18569252
- [Background] Olgiati E, Russell C, Soto D, Malhotra P. Motivation and attention following hemispheric stroke. Prog Brain Res. 2016;229:343-366. doi: 10.1016/bs.pbr.2016.06.011. Epub 2016 Sep 16. PMID 27926447
- [Background] Oyake K, Suzuki M, Otaka Y, Tanaka S. Motivational Strategies for Stroke Rehabilitation: A Descriptive Cross-Sectional Study. Front Neurol. 2020 Jun 10;11:553. doi: 10.3389/fneur.2020.00553. eCollection 2020. PMID 32587572
- [Background] Raglio A, Zaliani A, Baiardi P, Bossi D, Sguazzin C, Capodaglio E, Imbriani C, Gontero G, Imbriani M. Active music therapy approach for stroke patients in the post-acute rehabilitation. Neurol Sci. 2017 May;38(5):893-897. doi: 10.1007/s10072-017-2827-7. Epub 2017 Jan 30. PMID 28138867
- [Background] Ripolles P, Rojo N, Grau-Sanchez J, Amengual JL, Camara E, Marco-Pallares J, Juncadella M, Vaquero L, Rubio F, Duarte E, Garrido C, Altenmuller E, Munte TF, Rodriguez-Fornells A. Music supported therapy promotes motor plasticity in individuals with chronic stroke. Brain Imaging Behav. 2016 Dec;10(4):1289-1307. doi: 10.1007/s11682-015-9498-x. PMID 26707190
- [Background] Schaefer RS. Auditory rhythmic cueing in movement rehabilitation: findings and possible mechanisms. Philos Trans R Soc Lond B Biol Sci. 2014 Dec 19;369(1658):20130402. doi: 10.1098/rstb.2013.0402. PMID 25385780
- [Background] Schneider S, Schonle PW, Altenmuller E, Munte TF. Using musical instruments to improve motor skill recovery following a stroke. J Neurol. 2007 Oct;254(10):1339-46. doi: 10.1007/s00415-006-0523-2. Epub 2007 Jan 27. PMID 17260171
- [Background] Stone SP, Ali B, Auberleek I, Thompsell A, Young A. The Barthel index in clinical practice: use on a rehabilitation ward for elderly people. J R Coll Physicians Lond. 1994 Sep-Oct;28(5):419-23. PMID 7807430
- [Background] Street AJ, Magee WL, Odell-Miller H, Bateman A, Fachner JC. Home-based neurologic music therapy for upper limb rehabilitation with stroke patients at community rehabilitation stage-a feasibility study protocol. Front Hum Neurosci. 2015 Sep 23;9:480. doi: 10.3389/fnhum.2015.00480. eCollection 2015. PMID 26441586
- [Background] Street, A., Fachner, J. & Magee, W. (2019) Upper limb rehabilitation in chronic stroke using neurologic music therapy: Two contrasting case studies to inform on treatment delivery and patient suitability, Nordic Journal of Music Therapy, 28:5, 382-404, DOI: 10.1080/08098131.2019.1606848
- [Background] Thaut, M. H., & Hoemberg, V. (Eds.). (2014). Handbook of neurologic music therapy. Oxford University Press.
- [Background] Tong Y, Forreider B, Sun X, Geng X, Zhang W, Du H, Zhang T, Ding Y. Music-supported therapy (MST) in improving post-stroke patients' upper-limb motor function: a randomised controlled pilot study. Neurol Res. 2015 May;37(5):434-40. doi: 10.1179/1743132815Y.0000000034. Epub 2015 Apr 27. PMID 25916420
- [Background] Verrienti G, Raccagni C, Lombardozzi G, De Bartolo D, Iosa M. Motivation as a Measurable Outcome in Stroke Rehabilitation: A Systematic Review of the Literature. Int J Environ Res Public Health. 2023 Feb 26;20(5):4187. doi: 10.3390/ijerph20054187. PMID 36901206
- [Background] van Alphen R, Stams GJJM, Hakvoort L. Musical Attention Control Training for Psychotic Psychiatric Patients: An Experimental Pilot Study in a Forensic Psychiatric Hospital. Front Neurosci. 2019 Jun 7;13:570. doi: 10.3389/fnins.2019.00570. eCollection 2019. PMID 31231183